CLINICAL TRIAL: NCT04607967
Title: Efficacy of High Flow Nasal Oxygen Therapy Started in the Emergency Room Versus Conventional Oxygen Therapy in Patients With Acute Hypoxemic Respiratory Distress
Brief Title: HFNO or Conventional Oxygen Therapy for Patients With Acute Hypoxemic Respiratory Distress
Acronym: HIFLOWED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); centre Hospitalier Intercommunal de Vesoul (Unknown); Centre Hospitalier Universitaire de Saint Louis APHP (Unknown); Poitiers University Hospital (Other); University Hospital, Clermont-Ferrand (Other); Rennes University Hospital (Other); Centre Hospitalier of Chartres (Other); University Hospital, Toulouse (Other); University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/472
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-04

CONDITIONS: Acute Hypoxemic Respiratory Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional oxygen-therapy (study group "CO") (No Intervention): Patients randomized in the "Conventional Oxygen" group will be treated according to the national and international recommendations with a conventional oxygen-therapy device (nasal cannula or nasal-oral mask).
  Treatment failure will be evaluated after 4 hours by the need for a therapeutic escalation.
- High Flow Nasal Oxygen (study group "HNFO") (Experimental): Patients randomized in the "HNFO" group will be treated according to the CE Marking with the high flow nasal oxygen device.
  Treatment failure will be evaluated after 4 hours by the need for a therapeutic escalation.
  Interventions: Device: High Flow Nasal Oxygen

INTERVENTIONS:
Device: High Flow Nasal Oxygen — Study participants are suffering from an acute hypoxemic respiratory distress. They have to be treated with oxygen-therapy that could be administered using a conventional oxygen device (study group "CO") or High Flow Nasal Oxygen (study group "HNFO"). During the first 60 minutes following patients admission, patients will be randomized to one of the two study groups. In both groups, the failure of the treatment will be evaluated by the need for a therapeutic escalation fours hours after the treatment initiation.
  Other Names: HNFO (High Flow Nasal Oxygen)
  Arms: High Flow Nasal Oxygen (study group "HNFO")

SUMMARY:
A quarter of the patients admitted to the Shock Room or Resuscitation Room of an Emergency Department (ED) are admitted for severe hypoxemia resulting from acute respiratory distress. Like all life-threatening conditions, acute respiratory distress (ARD) requires a rapid identification and a prompt implementation of effective resuscitation measures.

Oxygen treatment, first described in 1890, remains one of the most important discoveries in medicine. The purpose of oxygenation is to alleviate respiratory failure and to restore a satisfactory hematosis. The choice of the oxygen delivery device is based on the severity of the hypoxemia, the underlying physiological problems, the type of dyspnea and the patient's tolerance to the device. The most commonly used devices are nasal cannula, face mask and high-concentration face mask (conventional oxygen therapy). High Flow Nasal Oxygen (HFNO) is now widely used as a complement to conventional oxygen therapy in the EDs.

HFNO ensures good clinical tolerance and better patient comfort (humidification and heating of inhaled gases...) than the other oxygen devices. The HFNO flow rate can go up to 60-70 L/min with an FIO2 (fraction of inspired oxygen inspired oxygen fraction) of 100% compared to a maximum output of 15 L/min with conventional oxygen-therapy.

Given the lack of data and clinical trials concerning the systematic use of HFNO in EDs in cases of severe hypoxemia, a prospective study is essential. The purpose of this work is to evaluate the contribution of early administration of HFNO for patients with acute non-hypercapnic respiratory distress presenting in the ED, with the aim of obtaining rapid correction of hematosis. The objective of this work is to compare Conventional Oxygen Therapy (CO) delivered by nasal cannula or nasal-oral mask at flow rates up to a maximum of 15 liters, to HFNO with the hypothesis that HFNO would reduce the need for ventilation therapy escalation. The other hypotheses concern the interest of the HFNO in reducing the use of intensive care hospitalization and thus the costs of treating these patients.

DETAILED DESCRIPTION:
Acute Respiratory Distress (ARD) is defined as the inability of a patient to maintain normal hematosis. A hematosis disorder is defined as an alteration of the blood gases with hypoxemia (partial pressure of oxygen (PaO2) less than 80 mm of mercury (mmHg) and transcutaneous O2 saturation (SpO2) less than 95%), associated or not with hypercapnia (partial pressure of carbon dioxide (PaCO2) > 45 mmHg) or hypocapnia depending on the cause of the acute respiratory failure. Compensation mechanisms include increased minute ventilation, increased ventilatory work and increased cardiac output. When these compensatory mechanisms are insufficient, acute respiratory distress occurs, along with signs of heart failure (acute cor pulmonale) and neuropsychic disorders.

Without care, a potentially fatal respiratory decompensation may occur. ARD can be hypercapnic. It's defined as a PaCO2 greater than 45 mm Hg associated with a drop in blood pH reflecting respiratory acidosis. Hypoxemic ARD is defined as a PaO2 of less than 60 mm Hg.

A quarter of the patients admitted to the Vital Emergency Room are admitted for severe hypoxemia resulting from acute respiratory distress.

Like all life-threatening conditions, acute respiratory distress (ARD) requires a rapid identification and a prompt implementation of effective resuscitation measures.

Oxygen treatment, first described in 1890, remains one of the most important discoveries in medicine. The purpose of oxygenation is to alleviate respiratory failure and to restore a satisfactory hematosis. Most experts stress the importance of having an SpO2 target of more than 90% in the majority of patients. While non-invasive ventilation (NIV) is the standard of care in the initial management of patients with hypercapnic acidosis, there are currently no recommendations for oxygen therapy in patients with acute hypoxic respiratory distress in the emergency department.

The choice of the oxygen delivery device is based on the severity of the hypoxemia, the underlying physiological problems, the type of dyspnea and the patient's tolerance to the device. The most commonly used devices are nasal cannula, face mask and high-concentration face mask. They offer several Oxygen Inspired Fraction (fraction of O2 in the gas mixture breathed, FiO2) depending on the oxygen flow rate instituted.

High Flow Nasal Oxygen (HFNO) is used as a complement to conventional oxygen therapy in emergency departments in general and in particular in the different emergency departments participating in our study. HFNO is used in hypoxemic respiratory insufficiency according to the national and international recommendations.

HFNO makes it possible to administer a much higher flow of oxygen than with the usual hospital and prehospital flow meters. This flow rate can go up to 60-70 L/min with an FIO2 of 100%. This high flow rate allows to generate low levels of positive pressure in the upper airways and to adapt the FIO2 delivered up to 100% notably thanks to dedicated nasal cannulas. HFNO ensures good clinical tolerance and better patient comfort (humidification and heating of inhaled gases ...) than the other oxygen devices. Its use was initially developed in paediatric and neonatal intensive care units. It was then gradually extended to "adult" intensive care units and intensive care units in the treatment of hypoxemic, non-hypercapnic acute respiratory failure (ARF) with no indication for orotracheal intubation. The FLORALI study confirms its use as an alternative to conventional oxygen therapy in intensive care units. Its implementation, its efficacy (improvement of dyspnea, clinical respiratory signs and oxygenation parameters), its good tolerance and acceptability by the nursing staff, were recently demonstrated in an emergency department in 17 patients with hypoxic respiratory insufficiency. However, despite the increasing number of studies, methodologically heterogeneous and of insufficient statistical power, carried out on HFNO, these studies remain non-contributory with regard to the superiority of high nasal flow compared to conventional oxygen therapy. The gain of the HFNO strategy seems to be established for clinical ventilatory parameters and dyspnea level. However, the need for therapeutic escalation and mortality have not been precisely evaluated. On the other hand, there is very little information on the time required for the implementation of HFNO in the various studies carried out in patients. The available data indicate that the average time would usually be more than 90 minutes.

Given the lack of data and clinical trials concerning the systematic use of HFNO in emergency departments in cases of severe hypoxemia, a prospective study is essential. The purpose of this work is to evaluate the contribution of early administration of HFNO for patients with acute non-hypercapnic respiratory distress presenting in the emergency department, with the aim of obtaining rapid correction of hematosis. The objective of this work is to compare Conventional Oxygen Therapy (CO) delivered by nasal cannula or nasal-oral mask at flow rates up to a maximum of 15 liters to HFNO, with the hypothesis that HFNO would reduce the need for ventilation therapy escalation. The other hypotheses concern the interest of the HFNO in reducing the use of intensive care hospitalization and thus the costs of treating these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Admitted to the Emergency Department for acute respiratory distress :
* Respiratory rate ≥ at 25 cycles/min.
* And SpO2 ≤ at 95% without or with oxygen whatever the mode.
* And clinical signs of respiratory distress (pulling, thoraco-abdominal swinging).
* And PaO2/FIO2 ratio < 300mmHg.

Exclusion Criteria:

* Hypercapnic patients (PaCO2 > 45mmHg) with respiratory acidosis (pH<7.30).
* Indication for non-invasive ventilation or early invasive mechanical ventilation according to current scientific recommendations (acute pulmonary edema, Chronic obstructive pulmonary disease decompensation, or others).
* Dyspnea of traumatic origin.
* Traumatic pneumothorax.
* Hemodynamic instability (PAM<65mmHg).
* Patients treated with Mobile Emergency and Resuscitation Service (SMUR) who have already received cardiac or pulmonary treatment.
* Patients with cognitive deterioration (Glasgow score less than 13, dementia or mental failure that would prevent good cooperation).
* Patients with lesion(s) of the oro-nasal sphere contraindicated for the implementation of High Flow Nasal Oxygen Therapy.
* Subject unlikely to cooperate in the study and/or low cooperation anticipated by the investigator.
* Subject without health insurance.
* Pregnant woman.
* Subject being in the exclusion period of another study or included in the "national volunteer file".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2025-05-23 (Estimated); Study Completion 2025-06-23 (Estimated)

PRIMARY OUTCOMES:
Therapeutic escalation | 4 hours after treatment initiation
  The need for a therapeutic escalation will be searched 4 hours after treatment initiation (either Conventional Oxygen or High Flow Nasal Oxygen)

SECONDARY OUTCOMES:
Identification of possible early prognostic factors for HFNO failure, defined as the need for a therapeutic escalation, within 60 minutes after its initiation. | 60 minutes after treatment initiation
  Clinical criteria (respiratory rate, SpO2, signs of respiratory failure (pulling, laboured breathing), dyspnoea score measured by the modified Borg scale).
  Paraclinical criteria: PaO2/FIO2 ratio<300mmHg.
Assessment of the effectiveness of HNFO on patient outcomes (Total time of HNFO use in the ED, ED length of stay, length and type of hospitalization, and patient's status at 30-day (deceased, still hospitalized or discharged from the hospital).) | 30 days after treatment initiation
Etiology of dyspnea | 30 days after treatment initiation
  To describe the aetiology of dyspnoea (impairment of pulmonary neuromuscular function, secondary to chronic or acute obstructive pulmonary diseases, alveolar processes, vascular diseases, COVID, other).

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - University Hospital of Dijon, Dijon, Bourgogne-Franche-Comté
  - University Hospital of Besançon, Besançon, Franche Comté
  - Hospital of Chartres, Chartres
  - University Hospital of Clermont Ferrand, Clermont-Ferrand
  - Montpellier University Hospital, Montpellier
  - University Hospital of Lariboisière, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Rennes, Rennes
  - University Hospital of Toulouse, Toulouse
  - Hospital of Vesoul, Vesoul

IPD SHARING:
Plan to Share IPD: Undecided
The data in this study are not publicly available, but reasonable requests can be made to the corresponding author.

REFERENCES:
- [Derived] Pretalli JB, Parmentier AL, Mauny F, Desmettre T, Marjanovic N, Capellier G, Khoury A. Efficacy of high-flow nasal oxygen therapy started in the emergency room versus conventional oxygen therapy in patients with acute hypoxaemic respiratory distress: protocol for a French multicentric, prospective, open and randomised superiority study protocol (HIFLOWED). BMJ Open. 2024 Aug 19;14(8):e083262. doi: 10.1136/bmjopen-2023-083262. PMID 39160110